CLINICAL TRIAL: NCT05487599
Title: An Open-label, Dose-Finding, Phase 1/2 Study to Evaluate the Safety and Tolerability of a Single Intravenous Dose of LY3884961 in Patients With Peripheral Manifestations of Gaucher Disease (PROCEED)
Brief Title: A Clinical Trial of PR001 (LY3884961) in Patients With Peripheral Manifestations of Gaucher Disease (PROCEED)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prevail Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J3Z-MC-OJAE
Record Dates: First submitted 2022-06-01; First posted 2022-08-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Gaucher Disease; Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3884961 (Experimental): LY3884961 is an advanced therapy investigational medicinal product administered as a single intravenous infusion.
  Interventions: Genetic: LY3884961

INTERVENTIONS:
Genetic: LY3884961 — • LY3884961 is a replication-incompetent recombinant adeno-associated virus (AAV) vector. The vector is composed of a ss DNA genome packaged in an AAV-derived protein capsid.

SUMMARY:
Study J3Z-MC-OJAE is a Phase 1/2, multicenter, open-label, dose-finding study of LY3884961 evaluating the safety and tolerability in adults with peripheral manifestations of GD.

Up to 3 dose levels of LY3884961 will be assessed in 3 dose-finding cohorts of 3 patients. Following this, up to 6 patients may be enrolled in an expansion cohort.

For each enrolled patient, the study will be approximately 5 years in duration, including up to a 60-day screening period. During the first 18 months after dosing, subjects will be evaluated for the effects of LY3884961 on safety, tolerability, immunogenicity, biomarkers, and efficacy. Patients will be followed for an additional 42 months to monitor safety, immunogenicity, and selected biomarker and efficacy parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater or equal to 18 years at the time of informed consent.
2. Bi-allelic pathogenic GBA1 variants must be centrally confirmed.
3. On ERT or SRT for at least 2 years and on a stable, maximum tolerated dose, for at least 3 months prior to screening.
4. Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
5. Females and males will be eligible for this study. Men and women of childbearing potential must use a highly effective method of contraception consistently and correctly for the duration of the study, including the long-term follow-up.
6. Patients must agree to abstain from blood, tissue and organ donation; and must agree to abstain from tissue and organ donation for the duration of the study, including long-term follow-up.

Exclusion Criteria:

1. Clinically significant neurological signs and symptoms and/or behavioral disturbances.
2. Active and progressive bone disease expected to require surgical treatment in the next 6 months.
3. History of total splenectomy or planned total splenectomy during the first 18 months of the study. (Partial splenectomy not exclusionary).
4. Splenomegaly > 10 MN as evaluated by centrally read abdominal magnetic resonance imaging (MRI)
5. Evidence of clinically significant liver disease, fragile liver, or history of exposure to hepatotoxins.
6. Thrombocytopenia with platelet count < 40 × 10^3 per μL.
7. Severe hyperlipidemia (triglycerides > 1,000 mg/dL).
8. Current diagnosis of unstable or clinically significant cardiovascular conditions based on Investigator assessment.
9. History of certain cancers within 5 years of Screening.
10. Concomitant disease, condition or treatment which, in the opinion of the Investigator, would pose an unacceptable risk to the patient or interfere with the patient's ability to comply with study procedures or interfere with the conduct of the study.
11. Women of childbearing potential, pregnant (i.e., positive serum pregnancy result at Screening and/or Check-in) or breastfeeding or intending to become pregnant during the course of the trial.
12. Use of any GD-related chaperone therapy within 4 weeks prior to Screening or expected need to initiate chaperone therapy during at least the first 18 months of the study.
13. Any type of prior gene or cell therapy.
14. Use of systemic immunosuppressant or steroid therapy other than protocol-specified immunosuppression.
15. Participation in another therapeutic investigational drug or device study within 3 months or 5 half-lives of the study agent, whichever is longer.
16. Have an anti-AAV9 antibody titer of >1:40 as determined by central laboratory.
17. Clinically significant abnormalities in laboratory test results at Screening.
18. Have any contraindications for MRI, including claustrophobia or the presence of contraindicated metal (ferromagnetic)implants/cardiac pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2031-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | 5 years
  Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) with AE's graded as mild, moderate, or severe.

SECONDARY OUTCOMES:
Spleen volume | 5 years
  Change and percent change from baseline
Platelet count | 5 years
  Change from baseline
GCase levels | 5 years
  Change from baseline
GlcSph levels | 5 years
  Change from baseline
Discontinuation of enzyme replacement therapy (ERT)/substrate reduction therapy (SRT) | 5 years
  Time from dosing to discontinuation of ERT/SRT
Re-initiation of ERT/SRT (if necessary) | 5 years
  Time to development of criteria requiring re-initiation of ERT/SRT (if necessary)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Neuhaus, DO, Study Director — Prevail Therapeutics, a wholly owned subsidiary of Eli Lilly and Company
Locations (8):
- United States (3):
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Duke University Health System, Durham, North Carolina
  - Lysosomal & Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Westmead Hospital-Cnr Hawkesbury and Darcy Rds, Westmead, New South Wales, Australia
- Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil
- SphinCS Clinical Science for LSD, Höchheim, Germany
- Hospital Quironsalud Zaragoza, Paseo Mariano Renovales Sn, Zaragoza, Spain
- Royal Free Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No